CLINICAL TRIAL: NCT07140640
Title: Effect of a 20% Reduction in Hyperbaric Bupivacaine Dose on High Spinal Block Incidence in Cesarean Delivery: A Risk-Stratified Randomized Controlled Trial.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Eman Mahmoud, Resident Doctor, Aswan University
Allocation: Not Applicable | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1084-3-25
Record Dates: First submitted 2025-08-22; First posted 2025-08-25 (Actual); Last update posted 2025-08-25 (Actual); Status verified 2025-04

CONDITIONS: Cesarean Section Complications
Keywords: cesarean-20% hyperbaric bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard dose of Hyberbaric Bupivacaine in Elective cesarean section (Active Comparator): 1- Standard dose group: receiving the typical dose of hyperbaric bupivacaine (12.5 mg hyperbaric bupivacaine + 25 mcg fentanyl).
  Interventions: Drug: Hyperbaric Bupivacaine HCl 0.5% 12.5 mg
- Reduced dose group in Elective cesarean section (Active Comparator): 2- Reduced dose group: receiving a20% reduced dose of hyperbaric bupivacaine (10 mg hyperbaric bupivacaine + 25 mcg fentanyl).
  Interventions: Drug: Hyperbaric Bupivacaine HCl 0.5% 10 mg

INTERVENTIONS:
Drug: Hyperbaric Bupivacaine HCl 0.5% 12.5 mg — 1- Standard dose group: receiving the typical dose of hyperbaric bupivacaine (12.5 mg hyperbaric bupivacaine + 25 mcg fentanyl).
  Other Names: Standard dose of hyperbaric bupivacaine
  Arms: Standard dose of Hyberbaric Bupivacaine in Elective cesarean section
Drug: Hyperbaric Bupivacaine HCl 0.5% 10 mg — 2- Reduced dose group: receiving a20% reduced dose of hyperbaric bupivacaine (10 mg hyperbaric bupivacaine + 25 mcg fentanyl).
  Other Names: 20% reduced dose of hyperbaric bupivacaine
  Arms: Reduced dose group in Elective cesarean section

SUMMARY:
Effect of a 20% Reduction in Hyperbaric Bupivacaine Dose on High Spinal Block Incidence in Cesarean Delivery: A Risk-Stratified Randomized Controlled Trial.

DETAILED DESCRIPTION:
This an interventional study comparing effect of Standard dose of Hyperbaric bupivacaine with 20% reduction of dose of Hyperbaric Bupivacaine in Elective Cesarean Delivery.

First, we determaine if the patient ( low - moderate - high ) risk to High spinal complication or not according to : Age-weight-BMI-Height.

Then , Randomly we gave the patients " Full dose of Hyperbaric Bupivacaine OR 20% reduction of hyperbric Bupivacaine " in spinal anaethsia .

Post anesthesia evaluation:

to assess incomplete sensory and/or motor blockade after spinal anesthesia for cesarean section is the Bromage Scale for motor blockade and a sensory block assessment using pinprick or cold sensation.

1. Bromage Scale for Motor Blockade:

   This scale assesses the degree of motor block in the lower limbs:
   * Grade 0: No paralysis, full flexion of knees and feet.
   * Grade 1: Inability to raise extended legs; can move knees and feet.
   * Grade 2: Inability to flex knees; can move feet.
   * Grade 3: Complete paralysis of the lower limbs.

   Incomplete motor blockade would typically be Bromage 1 or 2.
2. Sensory Block Assessment:

   * Sensory block is often assessed using a pinprick test or cold sensation (ice or alcohol swab).
   * Levels are recorded using dermatome levels (T10, T6, T4, etc.).
   * Incomplete sensory block means failure to achieve adequate sensory block (T4-T6 for cesarean section), requiring additional analgesia or conversion to general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* • Pregnant women aged 18-45 years.

  * ASA physical status II-III.

Exclusion Criteria:

* • Twin pregnancies.

  * Contraindications to spinal anesthesia (e.g., coagulopathy, infection).
  * Patients with incomplete preoperative data for risk stratification.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females planned for elective cesarean section
Enrollment: 333 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
1-Reduced Incidence of HSB | operation time
  1-reduced Incidence of HSB, defined as a sensory block level exceeding T4 within 15 minutes post-administration, accompanied by hemodynamic instability (e.g., hypotension >30% below baseline).
1-Reduced Incidence of HSB | first 20 minutes
  1-reduced Incidence of HSB, defined as a sensory block level exceeding T4 within 15 minutes post-administration, accompanied by hemodynamic instability (e.g., hypotension >30% below baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Mohamdy Eldemerdash, consultant, Study Director — Aswan University
Locations (1):
- Aswan university, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benjhawaleemas P, Sakolnagara BBN, Tanasansuttiporn J, Chatmongkolchart S, Oofuvong M. Risk prediction score for high spinal block in patients undergoing cesarean delivery: a retrospective cohort study. BMC Anesthesiol. 2024 Nov 11;24(1):406. doi: 10.1186/s12871-024-02799-w. PMID 39528929
- See also: Risk prediction score for high spinal block in patients undergoing cesarean delivery: a retrospective cohort study — https://pubmed.ncbi.nlm.nih.gov/39528929/